CLINICAL TRIAL: NCT07378553
Title: Multiparametric Ultrafast Ultrasound Evaluation of Skeletal Muscle in Duchenne and Becker Muscular Dystrophies
Brief Title: Multiparametric Ultrafast Ultrasound Biomarkers for Duchenne and Becker Muscular Dystrophies
Acronym: INNOVAN
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: AGENCE NATIONALE DE RECHERCHE (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC25_0273; 2025-A01398-41 (Other: ANSM)
Record Dates: First submitted 2025-11-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Duchene Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Ultrasound Imaging; Ultrafast Ultrasound; Muscle
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Age-matched Controls: Age matched non-affected men, matched for men with Becker and Duchenne Muscular Dystrophies
- Boys/Men with Duchenne Muscular Dystrophy: This group will include ambulatory and non-ambulatory boys/men with Duchenne Muscular Dystrophy ranging from 5-30 years old.
- Boys/Men with Becker Muscular Dystrophy: This group will include ambulatory and non-ambulatory men with Becker Muscular Dystrophy ranging from 5-60 years old.

SUMMARY:
The purpose of this research study is to determine the potential of a multiparametric ultrasound approach to non-invasively monitor disease progression and to serve as an objective outcome measure for future clinical trials in Duchenne and Becker Muscular Dystrophies.

The investigators will compare the muscles of ambulatory or non-ambulatory boys/men with Duchenne and Becker Dystrophies with muscles of healthy age-matched individuals of the same age and monitor disease progression in those with muscular dystrophies over a 12-month year period.

The ultrafast ultrasound technology used in this study allows the simultaneous assessment of muscle structure, mechanics and physiology, including stiffness, anisotropy, viscosity, intramuscular fat, muscle volume, and microvascular perfusion. The amount of muscle alteration measured will be related to performance in daily activities, such as walking and muscle strength, in order to identify sensitive and objective markers of disease progression.

DETAILED DESCRIPTION:
Duchenne and Becker muscular dystrophies (DMD/BMD) are the most common forms of muscular dystrophies, progressive muscle wasting diseases leading to weakness and devastating functional impairment. DMD is characterized by predominant involvement in skeletal, including respiratory, and cardiac muscles. Diagnosis is usually established at three to four years of age. Patients typically show muscle degeneration that worsens with age, leading to wheelchair dependency usually by the age of ten, assisted ventilation before the age of twenty, and premature death in the second to fourth decade. BMD shows a similar clinical phenotype but a later onset (approximately twelve years of age), a slower disease progression, delayed or no loss of ambulation, and variable involvement of the cardiac and respiratory systems. Considerable heterogeneity has been observed within and across the DMD/BMD phenotypes, which makes the design and analysis of clinical trials and prediction of the disease progression challenging.

Recent inconsistent results in DMD clinical development programs have also raised questions about the validity of the methods used to evaluate treatment efficacy. The number of potentially effective therapeutic approaches for DMD/BMD has rapidly increased over recent years, and thus the demand for validated outcome measures to demonstrate clinically meaningful therapeutic response over time in clinical trials (e.g., one year) is higher than ever. Regulatory agencies (e.g., FDA) have explicitly been encouraging the development of imaging biomarkers that may serve as surrogate markers of how patients will respond to investigational treatments in DMD/BMD.

This study aims to validate the potential of innovative ultrasound imaging methods, developed by our research consortium over recent years, as imaging tools to monitor disease progression and serve as a surrogate outcome measure for clinical trials in muscular dystrophies. Using cutting-edge ultrasound imaging techniques, including shear wave elastography, matrix approach, 3D freehand ultrasound, and power Doppler we will quantify much needed surrogate measures of muscle damage and progressive degeneration such as intramuscular fat content, fibrosis, muscle apoptosis and structural disorganization, inflammation, hypertrophy/atrophy, and intramuscular blood flow, in the lower and upper extremity muscles. An easy-to-apply multiparametric approach will be developed to assess the most important hallmarks of muscle degeneration associated with the most common and devastating muscular dystrophies.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for patients with Duchenne Muscular Dystrophy: Ambulatory and non-ambulatory males (ages 5-30 at baseline testing) previously diagnosed with Duchenne Muscular Dystrophy based on absence of dystrophin expression.
* Inclusion Criteria for patients with Becker Muscular Dystrophy: Ambulatory and non-ambulatory males (ages 5-60 at baseline testing) previously diagnosed with Becker Muscular Dystrophy based on genetically confirmed, reduced or dysfunctional dystrophin.
* Inclusion Criteria for Aged-matched controls: Ambulatory males (ages 5-60 years) without disease or injury to the lower and/or upper extremities

Exclusion Criteria:

* Exclusion Criteria for patients with Duchenne and Becker Muscular Dystrophies:

Inability to undergo static exam, missing measurement site (resection/amputation), neurocognitive impairment preventing informed consent

* Exclusion Criteria for Age-matched controls: Any condition affecting muscle metabolism/function, neuromuscular disease, or injury to the lower and/or upper extremities in the past 5 years

Ages: 5 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study Population
  This bicentric study will include 60 participants:
  18 male patients with Duchenne Muscular Dystrophy (DMD), aged 5 to 30 years (ambulant and non-ambulant),
  18 male patients with Becker Muscular Dystrophy (BMD), aged 5 to 60 years,
  and 24 healthy male subjects, aged 5 to 60 years, without neuromuscular disease or limb injury.
  All participants must have French social insurance coverage and provide informed consent (from parents or legal representatives for minors).
  Patients will be recruited mainly from the CHU de Nantes, the Institut de Myologie (Paris), and through the French Muscular Dystrophy Association (AFM-Téléthon). Healthy volunteers will be recruited from Nantes University staff, students, and their children.
  The inclusion of minors is necessary because Duchenne and Becker muscular dystrophies are X-linked genetic disorders diagnosed in childhood, and disease severity increases with age.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Baseline mechanical, structural, and physiological muscle ultrasound parameters | Baseline
  Assessment of muscle stiffness (kPa) in the lower extremity and/or upper extremity muscles across three participant groups
Baseline mechanical, structural, and physiological muscle ultrasound parameters | Baseline
  Assessment of anisotropy (a.u.) in the lower extremity and/or upper extremity muscles across three participant groups
Baseline mechanical, structural, and physiological muscle ultrasound parameters | Baseline
  Assessment of viscosity (Np/mm) in the lower extremity and/or upper extremity muscles across three participant groups
Baseline mechanical, structural, and physiological muscle ultrasound parameters | Baseline
  Assessment of nonlinear elastic parameters (kPa) in the lower extremity and/or upper extremity muscles across three participant groups
Baseline mechanical, structural, and physiological muscle ultrasound parameters | Baseline
  Assessment of intramuscular fat (m/s) in the lower extremity and/or upper extremity muscles across three participant groups
Baseline mechanical, structural, and physiological muscle ultrasound parameters | Baseline
  Assessment of intramuscular blood flow (%) in the lower extremity and/or upper extremity muscles across three participant groups

SECONDARY OUTCOMES:
Change from baseline in mechanical, structural, and physiological muscle ultrasound parameters | 12 months
  Assessment of muscle stiffness (kPa) in the lower extremity and/or upper extremity muscles across three participant groups
Change from baseline in mechanical, structural, and physiological muscle ultrasound parameters | 12 months
  Assessment of anisotropy (a.u.) in the lower extremity and/or upper extremity muscles across three participant groups
Change from baseline in mechanical, structural, and physiological muscle ultrasound parameters | 12 months
  Assessment of viscosity (Np/mm) in the lower extremity and/or upper extremity muscles across three participant groups
Change from baseline in mechanical, structural, and physiological muscle ultrasound parameters | 12 months
  Assessment of nonlinear elastic parameters (kPa) in the lower extremity and/or upper extremity muscles across three participant groups
Change from baseline in mechanical, structural, and physiological muscle ultrasound parameters | 12 months
  Assessment of intramuscular fat (m/s) in the lower extremity and/or upper extremity muscles across three participant groups
Change from baseline in mechanical, structural, and physiological muscle ultrasound parameters | 12 months
  Assessment of intramuscular blood flow (%) in the lower extremity and/or upper extremity muscles across three participant groups
Muscle function | Baseline and changes from baseline in at 12 months
  Muscle strength will be evaluated by dynamometry
Functional outcomes | Baseline and changes from baseline at 12 months
  10-Meter Walk Test in DMD and BMD participants
Functional outcomes | Baseline and changes from baseline at 12 months
  NorthStar Ambulatory Assessment performance in DMD and BMD participants
Correlations between ultrasound measures, muscle function and functional outcomes | Through study completion, 12 months
  In both BMD and DMD, the correlation between each ultrasound imaging parameter [muscle stiffness (kPa), anisotropy (a.u.), viscosity (Np/mm), nonlinear elastic parameters (kPa), intramuscular fat (m/s), muscle volume (ml), and intramuscular blood flow (%)] and all functional endpoints [NorthStar Ambulatory Assessment, 10-Meter Walk Test] will be determined, as well as the ability of ultrasound measures to predict future change and loss in function.